CLINICAL TRIAL: NCT02493205
Title: The Holding Area LINQ Trial is a Prospective, Non-randomized, Single Center Post-market Clinical Trial Designed to Occur in the Holding Area of a Hospital Operating Room or Cardiac Catheterization/Electrophysiology Laboratory
Brief Title: The Holding Area LINQ (Reveal LINQ Insertable Cardiac Monitor) Trial is a Prospective, Non-randomized, Single Center Post-market Clinical Trial
Acronym: HALT
Status: Completed | Type: Observational
Sponsor: Holy Cross Hospital, Florida (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Wilson Burke, Clinical Research Manager, Holy Cross Hospital, Florida
Other Study IDs: 201501RANA
Record Dates: First submitted 2015-06-30; First posted 2015-07-09 (Estimated); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
Keywords: Implantable Cardiac Monitor; Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Holding Area LINQ Trial is a clinical trial designed to compare the benefits in conducting impant procedures in the holding area of a hospital operating room vs cardiac catheterization/electrophysiology laboratory.

DETAILED DESCRIPTION:
The Holding Area LINQ Trial is a prospective, non-randomized, single center post-market clinical trial designed to occur in the holding area of a hospital operating room or cardiac catheterization/electrophysiology laboratory. The primary objective is to characterize the rate of procedure-related complications within 90 days of the implant procedure which require resolution by surgical intervention. Twenty (20) patients with established clinical indications for the LINQ ICM (Reveal LINQ Insertable Cardiac Monitor) will be implanted using standard of care techniques and procedures. Implants will be required to take place in a hospital holding area rather than the traditional facility locations such as the hospital operating room, cardiac catheterization lab, or electrophysiology lab. A physical description of the holding area is a small patient examination room separated from other patient exam bay by walls and a door. There is a sink in the patient exam room, laminate flooring, ceiling A/C vent, wall mounted Hemodynamic monitoring equipment, and wall mounted oxygen/suction lines. Patient sedation will be limited to local anesthetics and/or oral anti-anxiety medications. Intravenous access will be obtained only for emergency resuscitative measures. Due to the low complication rate for this type of implant and practical limitations on the sample size, there are no formal hypotheses tested in this trial. This study will characterize all procedure-related adverse events that occur within 90 days of the implant procedure. Data will be collected at implant, 7-10 day post-op visit, and 90-day post-implant visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is indicated for continuous arrhythmia monitoring with an Implantable Cardiac Monitor
2. Patient is willing to undergo implant in holding area setting with only local anesthetic and/or oral anti-anxiety medications for sedation (2 mg of Valium or Ativan) at patient request.
3. Patient is 18 years of age or older.
4. Patient is willing to provide informed consent and authorize disclosure of personal health information in accordance with state and national regulations.

Exclusion Criteria:

1. Patient has reduced immune function or is otherwise at high risk for infection
2. Patient has had a recent (within 30 days) or otherwise unresolved infection.
3. Patient is implanted or indicated for implant with a pacemaker, Implantable Cardiac Device (ICD), Cardiac Resyncronization Therapy (CRT) or hemodynamic monitoring system.
4. Patient is participating in another clinical trial that may have an impact on the trial endpoints.
5. Patient has a super-therapeutic INR > 3.0.
6. Patient considered by Principal Investigator and/or sub-investigator to be inappropriate for the trial for any reason.
7. Patient's life expectancy is less than 1 year.
8. Patient is pregnant.
9. Patient has an unusual thoracic anatomy or scarring at the implant site which may adversely affect the success of the implant procedure.
10. Inability to comply with planned trial procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 and older indicated for continuous arrhythmia monitoring with an Implantable Cardiac Monitor
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Rate of procedure-related complications within 90 days of implant which require resolution by surgical intervention. | 90 days post-implant.
  -For this study there is no formal hypothesis or performance criterion tested for this objective. Instead, the rate of these complications will be characterized by computing a point estimate and one-sided upper 95% confidence interval for the rate of procedure-related complications requiring surgical intervention 90 days post-implant-

SECONDARY OUTCOMES:
Cost-effectiveness for LINQ ICM holding area implants. | 90 days Post Implant
  Procedure duration as well as the types of personnel and resources needed for LINQ implant will be collected on the implant case report form. This information will be summarized using summary statistics and/or graphical methods.
Device functionality post-implant through patient trial exit visit. | 90 Days Post Implant
  Device functionality post-implant will be characterized by collecting R-wave amplitudes on the day of implant and at the 90-day follow-up visit. Following each implant, R-wave amplitude will be collected and recorded on the Implant e-CRF. In addition, R-wave amplitude will be collected and recorded at the 90-day follow-up visit or at an unscheduled visit should the patient exit the study prior to the 90-day follow-up visit. Summary statistics and/or graphical methods will be used to summarize the R-wave amplitude.
Resource utilization for LINQ ICM holding area implants. | 90 Days Post Implant
  Procedure duration as well as the types of personnel and resources needed for LINQ implant will be collected on the implant case report form. This information will be summarized using summary statistics and/or graphical methods.
Procedures utilized during LINQ ICM holding area implants. | 90 Days Post Implant
  Procedure duration as well as the types of personnel and resources needed for LINQ implant will be collected on the implant case report form. This information will be summarized using summary statistics and/or graphical methods.
Techniques utilized during LINQ ICM holding area implants. | 90 Days Post Implant
  Procedure duration as well as the types of personnel and resources needed for LINQ implant will be collected on the implant case report form. This information will be summarized using summary statistics and/or graphical methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Jim Moran Heart and Vascular Research Institute, Fort Lauderdale, Florida, United States